CLINICAL TRIAL: NCT03638544
Title: Effect of Wheat Bread and Pasta With Reduced Content of Gluten on Patients With Irritable Bowel Syndrome: Randomized Controlled Cross Over Study
Brief Title: Reduced Content of Gluten Diet on Patients With Irritable Bowel Syndrome (Pro.Ali.Fun.)
Acronym: PROALIFUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Prof, University of Bari
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PROALIFUN
Record Dates: First submitted 2018-07-11; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Irritable Bowel Syndrome; Gluten Sensitivity
MeSH Terms: conditions — Irritable Bowel Syndrome; Celiac Disease

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled Gluten Sensitivity
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced Gluten-Normal Gluten (Active Comparator)
  Interventions: Dietary Supplement: Reduced gluten bread and Pasta compared o normal gluten bread and Pasta
- Normal Gluten-Reduced Gluten (Active Comparator)
  Interventions: Dietary Supplement: Reduced gluten bread and Pasta compared o normal gluten bread and Pasta

INTERVENTIONS:
Dietary Supplement: Reduced gluten bread and Pasta compared o normal gluten bread and Pasta — Pasta with low gluten (50% of the normal) content achieved by optimization of techological parameters such as dough yield, time of fermentation and concentration of fungal proteases The gluten reduction is obtained without any other intervention of wheat breeding or the endogenous proteolytic enzymes of flours.

SUMMARY:
This study aim to manufacture bread and pasta with an reduced content of gluten and to assess the impact of reducing the daily intake of gluten by 50% in irritable bowel syndrome (IBS) patients. Fungal proteases and selected sourdough lactic acid bacteria will be used for making wheat bread and pasta with a reduced content of gluten (RG) (-50% of traditional products). From a technological point of view, the chemical, structural and sensory features of the RG products approached those of the bread and pasta made with normal level of gluten. The efficacy and safety of new products will be compared to traditional bread and pasta by using a double blind randomized, crossover-controlled trial in IBS patients with persistent gastrointestinal symptoms. Patients will follow two weeks of a GFD diet containing RG bread and pasta and two weeks of GFD diet containing Normal Gluten bread and pasta Symptoms severity will be assessed by Irritable Bowel Syndrome Severity Score (IBS-SS), Visual Analogue Scale (VAS), Hospital Anxiety and Depression Scale (HADS) and Irritable Bowel Syndrome Quality of Life (IBS-QoL).

ELIGIBILITY:
Inclusion Criteria:

1. age above 18 years;
2. having bowel symptoms (altered bowel habit, lower abdominal pain, bloating, or distention suggestive of IBS), as determined by Rome III criteria.
3. Previous exclusion of CD and wheat allergy

Exclusion Criteria:

1. previous GI malignancy and/or surgery;
2. clinically significant cardiovascular, respiratory, endocrine, renal, hematologic or hepatic disease.
3. other clinically significant medical condition; pregnancy or lactation; alcohol abuse; drug addiction; severe neurologic or psychiatric disorders; long-term use of corticosteroids or anti-inflammatory drugs
4. participation in another clinical trial within 6 months before the onset of this trial.

   -

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Severity of IBS symptoms measured by Irritable Bowel Syndrome-Severity Score (IBS-SS) | two weeks of each different diet interspersed by one week of wash out. The questionnaire will be completed ones a week.
  Change in IBS Severity Score (IBS-SS) between reduced gluten content diet and standard gluten content diet. Mild, moderate and severe cases were indicated by scores of 75 to 175, 175 to 300 and "300 respectively. Mild, moderate and severe cases are indicated by scores of 75 to 175, 175 to 300, and >300, respectively.
Change of IBS severity measured by Visual analogue scale (VAS) | Two weeks of each different diet interspersed by one week of wash out. The scale will be completed ones a day.
  Change of severity of IBS symptoms measured by Visual analogue scale (VAS) between reduced gluten content diet and standard gluten content diet. The 0-10 mm VAS scale (0 no pain, 10 worst possible pain) included a horizontal color gradient (green-red).

SECONDARY OUTCOMES:
Change of Quality of life scores | two weeks of each different diet interspersed by one week of wash out. The scale will be completed ones a week.
  Irritable Bowel Syndrome Quality of Life (IBS-QoL) between reduced gluten content diet and standard gluten content diet.

IPD SHARING:
Plan to Share IPD: No